CLINICAL TRIAL: NCT02086175
Title: A Phase 2 Clinical Trial of Rituxan and B-Glucan PGG in Relapsed Indolent Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: HiberCell, Inc. (Industry)
Responsible Party: Principal Investigator, Caron A. Jacobson, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-398
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Results first posted 2021-01-07 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Relapsed/Refractory Indolent B Cell Non-Hodgkin Lymphomas
Keywords: relapsed/refractory indolent B cell non-Hodgkin lymphomas
MeSH Terms: conditions — Recurrence | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imprime PGG and Rituximab (Experimental): The study drug, Imprime PGG, will be administered intravenously at a dose of 4mg/kg weekly for 4 weeks. Rituximab will be administered intravenously by institutional standards concurrently at a dose of 375mg/m2 weekly for 4 weeks. Response will be assessed with CT scans 10 weeks +/- 3 days following the completion of treatment
  Interventions: Drug: Imprime PGG; Drug: Rituximab

INTERVENTIONS:
Drug: Imprime PGG
Drug: Rituximab
  Other Names: IDEC-102; IDEC-C2B8; Rituxan; Mabthera

SUMMARY:
This research study is evaluating a drug combination called Imprime PGG and Rituximab as a possible treatment for relapsed/refractory indolent B cell non-Hodgkin lymphomas (NHL).

DETAILED DESCRIPTION:
After the screening procedures confirms eligibility:

Study Drugs: The participant will receive both Imprime PGG and rituximab weekly, for four weeks.

Clinical Exams: At the participant's weekly visit there will be have a physical exam and general health and specific questions about any problems they might be having and any medications the participant may be taking.

Scans (or Imaging tests):The Investigator will measure the participant's tumor 10 weeks after Week 4 of treatment by CT scan. Additional scans will be performed at 6 months and 12 months following the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Patients must have histologically determined indolent NHL that is relapsed or primary refractory after initial therapy. Indolent NHL includes the morphologic and clinical variants:

  * Follicular lymphoma, grades 1-3a
  * Marginal zone lymphoma (extranodal, nodal, or splenic)

    * All nodal marginal zone lymphomas are eligible
    * Extranodal marginal zone lymphomas of the stomach (gastric MALT lymphomas) may not be candidates for cure with antibiotics or local radiotherapy. Patients who have failed antibiotics or local therapy are eligible for the protocol as long as they have measurable disease and are naïve to chemotherapy and monoclonal antibody therapy.
    * Splenic marginal zone lymphoma patients may have received prior splenectomy as long as they have measurable disease and are naïve to chemotherapy and monoclonal antibody therapy.
  * Re-biopsy is not mandated at relapse unless there is clinical suspicion about an alternate diagnosis.
* Between 1-3 prior lines of chemoimmunotherapy and/or monotherapy with rituximab. Patients may not have had prior autologous or allogeneic stem cell transplantation.
* Measurable disease that has not been previously irradiated on CT scans of at least 2 cm, OR if the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation. Imaging must be completed no greater than 4 weeks prior to study enrollment.
* ECOG performance status 0-2 (Appendix B, Section 17.2)
* Absolute neutrophil count ≥1000 prior to treatment
* Oxygen saturation ≥ 90%, no more than 2 LPM oxygen
* Serum creatinine ≤ 1.5 X ULN
* AST ≤ 3 X ULN
* Total bilirubin ≤ 1.5 X ULN (unless there is lymphoma in the liver)
* Age ≥18 years
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 30 days of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.). Steroids for symptom palliation are allowed, but must be either discontinued or on stable doses at the time of initiation of protocol therapy.
* Patients may not be receiving any other investigational agents, or have received investigational agents within 4 weeks of beginning treatment.
* Patients who have previously received PGG-Betafectin (Betafectin®) or Imprime PGG.
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study.
* Patients with known leptomeningeal or brain metastases. Imaging or spinal fluid analysis to exclude CNS involvement is not required, unless there is clinical suspicion by the treating investigator.
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy or a known hypersensitivity to baker's yeast.
* Patients with known HIV infection or hepatitis B or C infection.HIV testing is not mandated and is to be performed at the discretion of the treating investigator.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Prior history of another malignancy (except for non-melanoma skin cancer or in situ cervical or breast cancer) unless disease free for at least three years. Patients with prostate cancer are allowed if PSA is less than 1.
* Patients should not receive immunization with attenuated live vaccine within one week of study entry or during study period.
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Women of child bearing potential (WOCBP) or male study participants of reproductive potential must agree to use double barrier birth control method of contraception during the course of the study treatment period and for 3 months after completing study treatment.

  -- WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who are not postmenopausal (no menses) for at least 12 consecutive months. WOCBP must have a negative urine or serum pregnancy test within 7 days prior to administration of treatment.
* History of noncompliance to medical regimens.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * New York Heart Association Class III or IV cardiac disease, including pre-existing clinically significant arrhythmia, congestive heart failure, or cardiomyopathy
  * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* Other uncontrolled intercurrent illness that would limit adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caron Jacobson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Imprime PGG and Rituximab: The study drug, Imprime PGG, will be administered intravenously at a dose of 4mg/kg weekly for 4 weeks. Rituximab will be administered intravenously by institutional standards concurrently at a dose of 375mg/m2 weekly for 4 weeks. Response will be assessed with CT scans 10 weeks +/- 3 days following the completion of treatment
  Imprime PGG
  Rituximab
Period: Overall Study
Arm/Group | Imprime PGG and Rituximab
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imprime PGG and Rituximab
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 12
Age, Continuous [Median (Full Range); unit: years] | 63 [40 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
ECOG Performance Status [Count of Participants; unit: Participants] — 0 = Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  1 = Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Participants
    0 - Fully Active | 18
    1 - Restricted | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate is percentage of participants with complete (CR) and partial (PR) responses as best response during treatment.
  CR:
  * Nodal Masses:
    1. For FDG-avid or PET positive prior to therapy; mass of any size permitted if PET negative
    2. For variably FDG-avid or PET negative; regression to normal size on CT.
  * Liver/Spleen:
  No palpable nodules
  -Bone Marrow Infiltrate cleared on repeat biopsy; if indeterminate by morphology, immunohistochemistry should be negative.
  PR:
  * Nodal Masses:
    * 50% decrease in SPD of up to 6 largest dominant masses; no increase in size of other nodes.
      1. FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site.
      2. Variably FDG-avid or PET negative; regression on CT.
  * Liver/Spleen:
    * 50% decrease in SPD of nodules; no increase in size of liver or spleen.
  * Bone Marrow:
  Irrelevant if positive prior to therapy; cell type should be specified.
Time Frame: Response assessed at week 14 of study calendar (10 weeks after the 4-week treatment regimen).
Population: All evaluated participants including two (2) non evaluable (NE) participants with partial or complete response (PR, CR)
Measure: Count of Participants; unit: Participants
Arm/Group | Imprime PGG and Rituximab
Number analyzed (Participants) | 25
Participants | 12
Statistical Analysis 1: Comparison: Imprime PGG and Rituximab; Patients will be accrued in a single stage design, with a goal accrual of 25 patients. Assuming a 30% response rate with rituximab alone, if the true but unknown rate of CR or PR is 50% with the addition of Imprime PGG, the probability of observing 11 or more patients with a response is 0.79 with 0.098 one-sided type-I error. Therefore a study with 25 patients, in which an observed response rate of 11/25 (44%) would be considered worthy of further consideration; Test type: Superiority; p = 0.044, Fisher Exact; percent = 48, 90% CI 2-sided [31 to 66]

2. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time from start of treatment to disease progression or death from any cause as estimated by Kaplan Meier methods. Patients who have not progressed and are alive are censored at the date the patient is known to be progression-free. Response is measure using the International Harmonization Project for Lymphoma criteria Cheson 2007, using CT scans of the chest, abdomen, and pelvis.
Time Frame: Patients were followed for a median (range) of 13.6 months (3-25).
Measure: Median (Full Range); unit: months
Arm/Group | Imprime PGG and Rituximab
Number analyzed (Participants) | 25
months | 14.4 [0 to 16]

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response DR is defined as the time from the date of first response (complete or partial) after treatment to the date of disease progression or death for any cause. Patients who are alive without progression are censored at the date the patient is last know to be progression-free.
Time Frame: Patients were followed for a median (range) of 13.6 months (3-25).
Measure: Median (Full Range); unit: months
Arm/Group | Imprime PGG and Rituximab
Number analyzed (Participants) | 25
months | 11.8 [0 to 12]

4. Secondary Outcome: Imprime PGG-bound Neutrophils Status by Response
Description: Imprime PGG-bound neutrophils analyzed using established methods (peripheral blood samples and post-treatment tumor samples to quantify the binding of Imprime PGG to neutrophils) by treatment response, best response.
Time Frame: Up to 14 weeks with a median (range of) 13 weeks (12-14).
Population: Imprime PGG-bound neutrophil status only available for this analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Imprime PGG and Rituximab
Number analyzed (Participants) | 22
Participants
  Imprime PGG-bound neutrophils: number analyzed (Participants) | 8
  Imprime PGG-bound neutrophils: Complete Response | 0
  Imprime PGG-bound neutrophils: Partial Response | 4
  Imprime PGG-bound neutrophils: Stable Disease | 4
  Imprime PGG-bound neutrophils: Progressive Disease | 0
  Non-bound neutrophils: number analyzed (Participants) | 14
  Non-bound neutrophils: Complete Response | 1
  Non-bound neutrophils: Partial Response | 5
  Non-bound neutrophils: Stable Disease | 4
  Non-bound neutrophils: Progressive Disease | 4

ADVERSE EVENTS:
Time Frame: Up to 66 weeks
Arm/Group | Imprime PGG and Rituximab
All-Cause Mortality (participants affected / at risk) | 2/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 12/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imprime PGG and Rituximab (N=25)
Infusion related reaction (General disorders) | 5 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Fatigue (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
White blood cell decreased (Investigations) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Joint pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT02086175/Prot_SAP_000.pdf